CLINICAL TRIAL: NCT03913780
Title: Impact of the Aerobic Exercise Versus Exercise of Force on the Hemodynamic, Lipidic, Anthropometric and Psychological Variables of Patients With Cardiac Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Tolteca (Other)
Responsible Party: Principal Investigator, Javier Eliecer Pereira Rodriguez, Physiotherapist, specialist in cardiopulmonary rehabilitation, magister in health sciences, university professor., University Tolteca
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: UTolteca
Record Dates: First submitted 2019-04-08; First posted 2019-04-12 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Heart Failure; Cardiac Failure
Keywords: Exercise; Force; Cardiac Rehabilitation; Rehabilitation; Heart Failure
MeSH Terms: conditions — Heart Failure; Motor Activity | interventions — Physical Conditioning, Human

STUDY DESIGN:
Intervention Model Description: 920 high-risk patients in cardiac rehabilitation, who after the exclusion criteria, 764 individuals were organized into 3 groups. This research for the group number 1 was retrospective with medical record and for groups 2 and 3 it was a randomized controlled trial with a basic probabilistic sampling by means of a table of random numbers, whose order was randomized through the Microsoft Excel 16.0 program, being the group experimental 1 at the end with 253 participants (aerobic exercise without strength training), 256 participants in experimental group 2 (aerobic exercise + strength training in the upper extremities) and control group with 255 (aerobic exercise + strength training for the lower extremities).
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Medical record) (Active Comparator): For group 1, participants do not have intervention as groups 2 and 3. This group consists of reviewing the medical history of the year 2000 to determine the variables of the study and then compare them with groups 2 and 3. This group of participants they were from the year 2000 and whose information will be strictly taken from their medical history was based on initial training with warm-up and walking, after that, aerobic training was performed from 50 to 70% of their maximum heart rate and they finished their session training with breathing exercises, coordination, balance and walking.
  Interventions: Other: Aerobic exercise more force
- Group 2: Aerobic exercise + Strength training in MMSS (Experimental): For group 2, participants begin their training with warm-up and walking, after that, performed aerobic exercise in endless band and elliptical bike more strength exercises for upper limbs with dumbbells, multi-strength equipment and Theraband.
  The prescription of aerobic exercise was given from 50 to 70% of your maximum heart rate and for strength, between 30% to 50% of 1 RM was determined, prolonging a percentage of heart rate that did not surpass 70% of the FCM nor the subjective uptake of physical effort to more than 6 on the modified Borg scale.
  Interventions: Other: Aerobic exercise more force
- Group 3: Aerobic exercise + Strength training in MMII (Experimental): For group 3, participants begin their training with warm-up and walking, after that, performed aerobic exercise in endless band and elliptical bike more the strength training for lower limbs with theraband, multi-strength equipment and exercises for activation of the sole-twin pump.
  The prescription of aerobic exercise was given from 50 to 70% of your maximum heart rate and for strength, between 30% to 50% of 1 RM was determined, prolonging a percentage of heart rate that did not surpass 70% of the FCM nor the subjective uptake of physical effort to more than 6 on the modified Borg scale.
  Interventions: Other: Aerobic exercise more force

INTERVENTIONS:
Other: Aerobic exercise more force — The work force for aerobic exercise is 50 to 70% of your maximum heart rate (HRM) achieved in the stress test according to the Naughton protocol. For strength, between 30% to 50% of 1 RM was determined, prolonging a percentage of heart rate that did not surpass 70% of the FCM nor the subjective uptake of physical effort to more than 6 on the modified Borg scale.
  Other Names: Physical training

SUMMARY:
Introduction and objectives: At the global level, cardiovascular diseases are the leading cause of mortality. Currently, rehabilitation programs are shown as an effective treatment to mitigate the effects of heart failure. The main objective is to compare the effects of aerobic exercise and strength in patients with heart failure after a cardiovascular rehabilitation program.

Methods and materials: Randomized controlled trial over a period of 3 years with patients with heart failure distributed in 3 groups (Aerobic exercise, aerobic exercise plus upper limb -MMSS- training, aerobic exercise plus training of lower limb -MMII-). Blood samples were taken to determine blood glucose levels and lipid profile. In addition, tests for aerobic capacity, maximum heart rate, anthropometry, depression, anxiety, clinical and hemodynamic parameters. The tests were performed before and after 24 training sessions, 60 min, 3 times a week for two months.

DETAILED DESCRIPTION:
MATERIALS AND METHODS

This research for the group number 1 was retrospective and for groups 2 and 3 it was a randomized controlled trial with a basic probabilistic sampling by means of a table of random numbers, whose order was randomized through the Microsoft Excel 16.0 program, being the group experimental 1 at the end with 253 participants (aerobic exercise without strength training), 256 participants in experimental group 2 (aerobic exercise + strength training in the upper extremities) and control group with 255 (aerobic exercise + strength training for the lower extremities). The present investigation was carried out in a period of 3 years (April 2016-2019) that contains the following attributes:

Characteristics of the participants The participants contained similar characteristics from the point of view of: ejection fraction, functional class, glucose, lipid profile, muscle percentage, fat and BMI (body mass index), abdominal circumference, overweight, obesity, prevalence of diabetes, arterial hypertension (HTA), kidney disease, cardiovascular risk factors and cardiovascular surgical procedure for their respective analysis. In addition, all participants presented "High risk" according to the stratification proposed by the American Association of Cardiopulmonary Rehabilitation. Highlighting that for group 1 their research methodology was retrospective through the collection of data from medical records of the year 2000 and groups 2 and 3 were interventions with methodology of randomized clinical trial between the years 2016 to 2019.

Criteria for inclusion in the study The patients had to be post-operative of cardiovascular surgery that go to a phase II cardiac rehabilitation program, which at the time had to sign an informed consent endorsed by the ethics and research committee of the institution. Likewise, it was necessary for participants to have heart failure with ejection fraction greater than 35%; do not have any inconvenience when doing the questionnaires, tests and measures that the investigation demands, and a commitment to go 3 times a week for RCV.

Exclusion criteria Patients who had severe pain in the lower limbs, unstable angina, heart rate >120 bpm (beats per minute) at rest, systolic blood pressure >190 mmHg, diastolic blood pressure >120 mmHg were discarded. Similarly, patients who had a positive contraindication item for cardiac rehabilitation were not admitted in the study. In addition, the participant had the option of being able to withdraw from the research when he wished or to show hemodynamic instability without improving during any test or during the intervention process.

Anthropometric measurement In all the participants the following data were obtained: Family and personal antecedents using a self-created questionnaire. Likewise, anthropometric measures (weight, height, body mass index, abdominal circumference, fat and muscle percentage) using standardized techniques in the Colombian population.

The weight, fat percentage and muscle, were obtained by using the digital scale previously calibrated and located on a flat and stable surface, using the indications in the user's manual. On the other hand, the size was obtained with the Kramer 2104 Adult Acrylic Wall Height Measurement, placing the patient standing, with the head in Frankfort plane and with the shoulders relaxed to avoid lordosis and MMII completely against the wall. Having said the above, with these variables the BMI was determined in kg/m-1.

Then, with a tape measure and a precision of 1mm, the abdominal circumference measurement was collected taking the anatomical referents described by Frisancho. The "Waist circumference cut points for the diagnosis of abdominal obesity in the Colombian population using bioimpedance as reference standard" were chosen as cutting points: in men 91cm and women 89cm.

Clinical and hemodynamic parameters After all the above procedures, the blood glucose levels were determined on the first and last day of your training session with an Acca-Chek® Perform glucometer following the technical specifications suggested by the manufacturer. The blood sample was taken between 7:00 and 8:00 a.m., after 8-10 hours of fasting. It should be added that the blood samples were collected in the hospital clinical laboratory to define cholesterol levels, triglycerides, low density lipoproteins (LDL) and high density lipoproteins (HDL). Each patient underwent a 2-D (two-dimensional) echocardiography before and after the cardiac rehabilitation program, to visualize the structures, the LVEF and analyze their mobility in real time. In this same evaluation, the functional class of each patient was identified according to the NYHA classification (New York Heart Association); which designates 4 classes (I, II, III and IV) based on the limitations of the patient's physical activity, caused by cardiac symptoms. Similarly, perceived dyspnea and effort were assessed using the modified Borg scale. The heart rate was detected by the Polar Multisport RS800CX system and the respiratory one, just as the systolic and diastolic blood pressure was obtained manually, while the oxygen saturation was obtained with a portable pulse oximeter (Nellcor Puritan Bennett).

Tests and questionnaires From the beginning, the patient underwent a medical assessment by the area of physiatry to understand the current state of the patient, sociodemographic, anthropometric and physiological characteristics. On the same day, tolerance to exercise was estimated by the 6-minute walk test, which was superimposed before and after 24 sessions of cardiac rehabilitation. The protocol of the 6-minute walk test was performed according to the ATS Statement: Guidelines for the six-minute walk test of the American Thoracic Society. On the other hand, to denote the initial weight of strength training for upper limbs (MMSS) and lower limbs (MMII), weights were used in a repetition with increase or decrease of the load of 2.5 to 8 lb, until achieving the maximum weight to lift. A maximum repetition (1RM) was considered appropriate with a full extension of the muscle group used, without muscle substitutions. After this evaluation day, the patient had to return to next day for an effort test according to the Naughton protocol, which is recommended in high-risk patients, with stages of 2 minutes. The patient was told that he should avoid smoking, drinking drinks or any type of drug or medication that could alter his vital signs or performance during the test.

Depression and anxiety The HADS questionnaire (Hospital Anxiety and Depression Scale) was used for anxiety and depression. Regarding anxiety, the questions are aimed at identifying if the user has been tense, worried or with some kind of fear. However, the questions of depression are aimed at identifying if the user shows disinterest in the activities of daily life, negativity about things and their attitude to be happy. At this point it is emphasized that the questionnaire was applied by two independent and blinded investigators (M. D-B and D. P-F); which delivered the questionnaires to two other investigators (R. P-R and L. C-P) for verification and analysis.

Blind methodology A simple blind clinical study was carried out, in which the patients were assessed by a non-research professional (physiatrist of the cardiac rehabilitation service), as well as blood tests. Afterwards, patients accessed a database in Microsoft Excel 16.0 exclusively with an identification number that allowed blinding of the investigators. Blindly, a first investigators (J. P-R) collected the database of 253 patients of total 564 intervened patients in cardiac rehabilitation in the year 2000 and provided the list to three blinded investigators (X. V-B, K. S-P and D. R-G) for form the group number 1. Likewise, the first investigators (J.P-R) captured the result of the assignment of the participants in the 2 cardiac rehabilitation groups and provided the list of experimental groups 2 and 3 to the blinded investigators P. P-R, D. P-F and M. D-B; R. P-R, C. Q-G and L. C-P; respectively.

For the groups 2 and 3, the researchers prepared the questionnaires and tests without them knowing the assignment of each patient. After the tests, participants were suggested to approach cardiac rehabilitation to let them know their schedule and start date to the training program. Ignoring the cardiopulmonary rehabilitators, after 24 training sessions according to the assigned group, they gave an accurate report on the physiological changes and behavior in each training session.

However, the initial tests until the end of the training program the investigators did not establish conversation about the topic with the participants or therapists. Exclusively the investigators J. P-R. held periodic meetings with the cardiopulmonary rehabilitators to be aware and harmonize the training of each group but not intimate with the participants.

After the training program, the tests and tests were carried out to the patients of each group to calculate the post-training changes. Taking into account the information collected pre- and post, the statistical analyzes for experimental group 1 were carried out by X. V-B, K. S-P and D. R-G; experimental group 2 for P. P-R, D. P-F and M. D-B and for the experimental group 3 the authors R. P-R, C. Q-G and L. C-P. Finally, once the different variables were studied in a blinded manner, all the authors were informed about the groups with their corresponding patients and results in order to produce the conclusions.

Intervention by group The cardiac rehabilitation program consisted of 24 sessions of 60 minutes a day (10 minutes of warm-up, 40 minutes of training and 10 minutes of cool down phase), 3 times a week, for two months. With regard to warming, it was based on mobilization exercises by muscle groups. Cool down phase was done with proprioception exercises, stretching coordination and breathing exercises.

Related to the 40 minutes of training, it was modified according to the assigned group, for the experimental group 1, it was supported only in aerobic exercise in endless band and elliptical bicycle (report by medical records). The patients of experimental group 2 performed aerobic exercise in endless band and elliptical bike as group 1 plus strength exercises for upper limbs with dumbbells, multi-strength equipment and Theraband. On the other hand, the training of the control group executed the same order of the experimental group 1 plus the strength training for lower limbs with theraband, multi-strength equipment and exercises for activation of the sole-twin pump.

The work force for aerobic exercise was 50 to 70% of your maximum heart rate (HRM) achieved in the stress test according to the Naughton protocol. For strength, between 30% to 50% of 1 RM was determined, prolonging a percentage of heart rate that did not surpass 70% of the FCM nor the subjective uptake of physical effort to more than 6 on the modified Borg scale.

ELIGIBILITY:
Inclusion Criteria:

* Participants in the cardiac rehabilitation program.
* To sign an informed consent endorsed by the ethics and research committee of the institution.
* Participants with heart failure with ejection fraction greater than 35%
* Participants do not have any inconvenience when doing the questionnaires, tests and measures that the investigation demands,
* Participants than will can to go 3 times a week for Cardiovascular rehabilitation.

Exclusion Criteria:

* Participants who had severe pain in the lower limbs.
* Unstable angina.
* Heart rate >120 bpm (beats per minute) at rest.
* Systolic blood pressure >190 mmHg.
* Diastolic blood pressure >120 mmHg.
* Participants who had a positive contraindication item for cardiac rehabilitation were not admitted in the study.
* Participants to show hemodynamic instability without improving during any test or during the intervention process.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 920 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Changes in ejection fraction after 24 training sessions (%) | After 2 month of training (24 training sessions)
  it is the most important measure of cardiac functioning. This value, expressed as a percentage, measures the decrease in the volume of the left ventricle of the heart in systole, with respect to the diastole. The normal values are higher than 45%
Changes in the Body weight after 24 training sessions (Kg) | After 2 month of training (24 training sessions)
  How much body weight (kg) pre and post intervention
Changes in the Body Mass Index after 24 training sessions (%) | After 2 month of training (24 training sessions)
  it is a mathematical reason that associates the mass and the size of an individual. it is also known as the Quetelet index. This result is determined by the formula of weight/square size.
Changes in the Abdominal circumference after 24 training sessions (cm) | After 2 month of training (24 training sessions)
  It is the measurement of the distance around the abdomen at a specific point. Abdominal circumference is used to diagnose and monitor abdominal obesity. The values are in centimeters and according to the population to be studied, the measurements must be less than 91cm for men and 89cm for women.
Changes in the Fat percentage after 24 training sessions (%) | After 2 month of training (24 training sessions)
  Percentage of body fat is considered a measure to determine the level of body fat and a high percentage is a risk factor that triggers multiple chronic diseases. This measure can be determined in many ways but in our study it was used by means of bioimpedance. The normal values for men and women depend on the age of the patients and the manufacturer of the scale.
Changes in the Muscle percentage after 24 training sessions (%) | After 2 month of training (24 training sessions)
  Muscle percentage is considered a measure to determine the level of muscle in the body and a low percentage is a risk factor that indicates sarcopenia and is associated with a decrease in quality of life. This measure can be determined in many ways but in our study it was used by means of bioimpedance. The normal values for men and women depend on the age of the patients and the manufacturer of the scale.
Changes in the levels of Depression and Anxiety after 24 training sessions | After 2 month of training (24 training sessions)
  Psychological alteration that can be determined by the "Hospital Anxiety and Depression Scale". This scale consists of a series of questions for depression and others for anxiety. The final grade is in the range of 1 to 10 and for the diagnosis of depression or anxiety the result must be greater than or equal to 8.
Changes in the levels of Total cholesterol after 24 training sessions (mg/dl) | After 2 month of training (24 training sessions)
  It is part of the measures to determine the lipid profile of a person and serves to determine different types of dyslipidemia. This item is obtained by means of a blood sample analyzed in a clinical laboratory and the result obtained by a professional for this purpose. Values above 200 mg/dl are indicative of a lipid alteration.
Changes in the levels of Triglycerides after 24 training sessions (mg/dl) | After 2 month of training (24 training sessions)
  It is part of the measures to determine the lipid profile of a person and serves to determine different types of dyslipidemia. This item is obtained by means of a blood sample analyzed in a clinical laboratory and the result obtained by a professional for this purpose. Values above 150 mg/dl are indicative of a lipid alteration.
Changes in the levels of LDL after 24 training sessions (mg/dl) | After 2 month of training (24 training sessions)
  It is part of the measures to determine the lipid profile of a person and serves to determine different types of dyslipidemia. This item is obtained by means of a blood sample analyzed in a clinical laboratory and the result obtained by a professional for this purpose. Values above 100 mg/dl are indicative of a lipid alteration.
Changes in the levels of HDL after 24 training sessions (mg/dl) | After 2 month of training (24 training sessions)
  It is part of the measures to determine the lipid profile of a person and serves to determine different types of dyslipidemia.This item is obtained by means of a blood sample analyzed in a clinical laboratory and the result obtained by a professional for this purpose. Values lower than 40 mg/dl are indicative of a lipid alteration.
Changes in the levels of Glucose after 24 training sessions (mg/dl) | After 2 month of training (24 training sessions)
  It is used to determine blood glucose levels and its high values are indicative for diabetes mellitus. This item is obtained by means of a blood sample analyzed in a clinical laboratory and the result obtained by a professional for this purpose. Values lower than 126 mg/dl are indicative of diabetes mellitus.
Changes in the Dyspnoea after 24 training sessions | After 2 month of training (24 training sessions)
  Dyspnea is a respiratory difficulty that usually translates into shortness of breath. Dyspnea can be determined using the original Borg scale (Score from 0 to 20) or modified (Score from 0 to 10), in which the higher the number indicated by the participant, the higher the degree of dyspnea.
Changes in the Fatigue after 24 training sessions | After 2 month of training (24 training sessions)
  It is a feeling of lack of energy, exhaustion or fatigue. The fatigue can be determined using the original Borg scale (Score from 0 to 20) or modified (Score from 0 to 10), in which the higher the number indicated by the participant, the higher the degree of fatigue.
Changes of the maximum heart rate in a effort test after 24 training sessions | After 2 month of training (24 training sessions)
  It is the maximum capacity that the heart has to contract and we determine it by means of an effort test. The Maximum heart rate can be determined by formula or in a effort test (In the present investigation) which consists in mounting the participant in an endless band with an inclination and speed determined according to the protocol for said test. The test is stopped when the participant. indicates that it can not be more or there are electrocardiographic alterations that indicate that it is the participant's maximum.

SECONDARY OUTCOMES:
Changes in the Estimated maximum oxygen volume after 24 training sessions (ml/kg/min) | After 2 month of training (24 training sessions)
  It is the maximum amount of oxygen that the body can absorb, transport and consume in a given time, is the blood that our body can transport and metabolize. To determine the Vo2 values, the 6-minute walking test is used and to determine the result of the test, formulas are used according to the meters traveled, age, sex, height and weight of the participant. The larger the meters traveled, the greater the vo2.
Changes in the unit of measurement of the metabolic index (METs) after 24 training sessions (ml/kg/min) | After 2 month of training (24 training sessions)
  It is the unit of measurement of the metabolic index (amount of energy consumed by an individual in a resting situation). To determine the METs values, the 6-minute walking test is used and to determine the result of the test, formulas are used according to the meters traveled, age, sex, height and weight of the participant. The larger the meters traveled, the greater the METs.
Changes in the Distance traveled after 24 training sessions (m) | After 2 month of training (24 training sessions)
  Distance traveled in this of 6 minute walk test. The larger the meters traveled, this will indicate better Vo2, METs and aerobic and physical capacity in the participant.

IPD SHARING:
Plan to Share IPD: No
Initially, it is an issue that depends on the hospital institution where the research was conducted due to the personal data of the patients and the confidentiality of the institution. Therefore, initially it would be to talk with the patients, the institution and all the researchers. Mainly with the clinic because it is a bit jealous with your information.